CLINICAL TRIAL: NCT06138236
Title: Comparison of ESWT and Collagen Hydrolyzed Peptides in the Treatment of Plantar Fascitiis
Brief Title: Plantar Fascitiis: Comparison of ESWT and Collagen Hydrolyzed Peptides
Acronym: PFESWTCP
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PFESWTCP
Record Dates: First submitted 2023-07-21; First posted 2023-11-18 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-07

CONDITIONS: Plantar Fascitis

STUDY DESIGN:
Intervention Model Description: Patients suffering from plantar fascitiis were randomized into three arms of treatment: Infiltration of collagen hydrolyzed peptides, ESWT and a combination of both treatments
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Infiltration (Experimental): 1. Infiltration of collagen hydrolyzed peptides
  Interventions: Drug: Collagen hydrolyzed peptides
- ESWT(Extracorporeal Shockwave Therapy) (Experimental): ESWT (Extracorporeal Shockwave Therapy)
  Interventions: Drug: Collagen hydrolyzed peptides
- Combination (Experimental): Combination of both treatments
  Interventions: Drug: Collagen hydrolyzed peptides

INTERVENTIONS:
Drug: Collagen hydrolyzed peptides — infiltration near the heal spur of 2ml of Arthrys
  Other Names: ESWT

SUMMARY:
Patients suffering from Plantar Fasciitis were randomized into three groups:

the first group underwent infiltration of Collagen Hydrolyzed Peptides, the second one underwent the ESWT treatment, the third one underwent a combination of the two treatments.

DETAILED DESCRIPTION:
Patients suffering from Plantar Fasciitis were randomized into three groups:

the first group underwent infiltration of Collagen Hydrolyzed Peptides, the second one underwent the ESWT treatment, the third one underwent a combination of the two treatments.

Aim of the study was to consider any difference in the outcome of the three groups of patients. The NRS and the AFAS score were considered for the outcome measurement.

ELIGIBILITY:
Inclusion Criteria:

Plantar fascitiis Aged between 18 and 80 years old

Exclusion Criteria:

* Previous surgery of the foot
* Contraindications to ESWT

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
VAS (Visuoanalogic scale) | Between recruitment and 30 days
  Visuoanalogic Scale during walking. Range 0 (No pain) -10 (maximum pain)
AFAS (American Foot and Ankle Score) is the American Foot and Ankle Scale | Between Recruitment and 15 days
  It is a measurement of active ROM and deambulation of the patient. Range 0 (no function) -100 (perfect function)
AFAS is American Foot and Ankle Scale | Between Recruitment and 30 days
  It is a measurement of active ROM and deambulation of the patient (Range 0-100)
AFAS is American Foot and Ankle Scale | Between Recruitment and 60 days
  It is a measurement of active ROM and deambulation of the patient (Range 0-100)

CONTACTS AND LOCATIONS:
Overall Officials: Silvana DE GIORGI, PI, Principal Investigator — University of Bari; Angela Notarnicola, AP, Study Chair — University of Bari
Locations (1):
- Angela Notarnicola, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lai TW, Ma HL, Lee MS, Chen PM, Ku MC. Ultrasonography and clinical outcome comparison of extracorporeal shock wave therapy and corticosteroid injections for chronic plantar fasciitis: A randomized controlled trial. J Musculoskelet Neuronal Interact. 2018 Mar 1;18(1):47-54. PMID 29504578
- [Result] Sun K, Zhou H, Jiang W. Extracorporeal shock wave therapy versus other therapeutic methods for chronic plantar fasciitis. Foot Ankle Surg. 2020 Jan;26(1):33-38. doi: 10.1016/j.fas.2018.11.002. Epub 2018 Nov 13. PMID 30502222
- [Result] Xu D, Jiang W, Huang D, Hu X, Wang Y, Li H, Zhou S, Gan K, Ma W. Comparison Between Extracorporeal Shock Wave Therapy and Local Corticosteroid Injection for Plantar Fasciitis. Foot Ankle Int. 2020 Feb;41(2):200-205. doi: 10.1177/1071100719891111. Epub 2019 Nov 19. PMID 31744313
- [Result] Melese H, Alamer A, Getie K, Nigussie F, Ayhualem S. Extracorporeal shock wave therapy on pain and foot functions in subjects with chronic plantar fasciitis: systematic review of randomized controlled trials. Disabil Rehabil. 2022 Sep;44(18):5007-5014. doi: 10.1080/09638288.2021.1928775. Epub 2021 May 26. PMID 34038642
- Available data/document: Study Protocol — https://www.sanita.puglia.it/web/policlinico-di-bari-ospedale-giovanni-xxiii/comitato-etico